CLINICAL TRIAL: NCT04665570
Title: Acarbose/Metformin Fixed Dose Combination: Treatment Patterns and Outcomes in Newly Diagnosed T2DM Patients in India
Brief Title: A Study to Learn More About How Acarbose and Metformin Work When Taken Together and How Safe They Are in Indian Patients Who Were Recently Diagnosed With Type 2 Diabetes (T2D)
Acronym: START-AM
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21455
Record Dates: First submitted 2020-10-23; First posted 2020-12-11 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose; Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment: The decision to prescribe Acarbose/Metformin fixed dose combination (FDC) will be solely at the discretion of the Investigator and in accordance with his/her experience. Patients can only be enrolled in the study if the decision to treat with Acarbose/Metformin fixed dose combination has been made by the treating physician in advance and independent of study inclusion.
  Interventions: Drug: BAY81-9783 (Acarbose/Metformin)

INTERVENTIONS:
Drug: BAY81-9783 (Acarbose/Metformin) — Tablet (FDC of 25/50mg acarbose + 500mg metformin), three times daily

SUMMARY:
The study drug, fixed dose combination of acarbose and metformin, have already been approved to take together as a treatment for type 2 diabetes (T2D). Sometimes, researchers continue studying a treatment after it has been approved to learn more about how doctors decide which treatment to give to patients. In this study, the researchers want to learn more about how acarbose and metformin work when taken together and if the patients have any medical problems.

The study will include patients with T2D that was diagnosed in the last 3 to 6 months. These patients will also have recently started treatment with acarbose and metformin. The study will include about 2,000 men and women in India who are at least 18 years old.

All of the patients will take fixed dose combination of acarbose and metformin tablets based on their doctor's instructions. They will then visit their study site 4 times over 6 months. At these visits, their doctors will ask them questions about how they are feeling and what medications they are taking. If require, the doctors will take blood samples to measure the patients' blood sugar levels as per routine practice. The doctors will also do physical examinations and check the patients' overall health.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed T2DM (diagnosed within last 3 to 6 months) patient eligible for dual therapy exhibiting HbA1c is ≥ 7.5% to 9.0% will be enrolled after decision to administer acarbose/metformin fixed dose combination for type-2 diabetes management has been made by the attending physician on the basis of best clinical practice and patient needs.
* Decision to initiate treatment with Acarbose/Metformin FDC was made as per Investigator's routine treatment practice
* Signed informed consent
* No participation in an investigational program with interventions outside of routine clinical practice
* No contra-indications according to the local prescribing information of GlucobayM

Exclusion Criteria:

* Patients receiving any other anti-diabetic medication than the study drug at the time of enrollment in the study will be excluded. However, during observation period, any additional anti-diabetics medication administered by the attending physician will be acceptable & recorded in case record form.
* Patients with type 1 diabetes
* Patients with HbA1c > 9%
* Patients who have serious infection, or have severe trauma
* Patients who are pregnant or breast-feeding, or have the potential to become pregnant and child bearing female patients who are not willing to use any birth control measures
* All contra-indications according to the local marketing authorization should be considered
* Patients with HbA1c with >9.0%: The target patient population is selected based on the AACE guideline recommendation to use combination therapy in case of higher glycaemia (HbA1c ≥7.5% - 9.0%) presented on diagnosis and also it is the common practice observed in India of using combination therapy in this group of patient as an initial therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male patients ≥ 18 years or older with a diagnosis of T2DM will be enrolled after the decision for treatment with acarbose/metformin FDC has been made by the Investigator. Patients who have been prescribed acarbose/metformin FDC for a medically appropriate use will be eligible to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2023-09-09 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Mean change in HbA1c | From baseline to end of week 24
  HbA1c: Glycated Hemoglobin

SECONDARY OUTCOMES:
Change in HbA1c | From baseline to end of week 12
Change in fasting blood glucose | From baseline to end of week 6, week 12, week 24
Change in postprandial glucose level | From baseline to end of week 6, week 12, week 24
Occurrence of Hypoglycemic events | From baseline up to 24 weeks
Severity of Hypoglycemic events | From baseline up to 24 weeks
Occurrence of Gastrointestinal intolerance | From baseline up to 24 weeks
Occurrence of other AEs relating to tolerability | From baseline up to 24 weeks
Change in patient tolerability to therapy | From baseline up to 24 weeks
Mean change in body weight | From baseline to end of week 12, week 24
Mean change in lipid profile | From baseline up to 24 weeks
Descriptive analysis of starting dose and final dosing | From baseline up to 24 weeks
Descriptive analysis of time taken for full dose titration | From baseline up to 24 weeks
Descriptive analysis of PPG recorded at each visit | From baseline up to 24 weeks
Descriptive analysis of FBG recorded at each visit | From baseline up to 24 weeks
Descriptive analysis of HbA1c recorded at each visit | From baseline up to 24 weeks
Descriptive analysis of body weight recorded at each visit | From baseline up to 24 weeks
Descriptive analysis of actual duration of treatment with acarbose/metformin FDC before addition of other anti-diabetes drugs | From baseline up to 24 weeks
Descriptive analysis of time of addition of the other anti-diabetes drug | From baseline up to 24 weeks
Descriptive analysis of reason of addition of the other anti-diabetes drug | From baseline up to 24 weeks
Descriptive analysis of reason for discontinuation of acarbose/metformin FDC treatment | From baseline up to 24 weeks
Descriptive analysis of adverse events (AEs) | From baseline up to 24 weeks
  AEs assessed and recorded by the physician on the AE report form attached to the case report form

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, India

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.